CLINICAL TRIAL: NCT03190148
Title: Explorative Study: Diagnosis and Medical Care of Disturbances of Glucose Metabolism in Pregnant Women With a History of Bariatric Surgery, Normal Weight and Obese Pregnant Women
Brief Title: Glucose Metabolism in Pregnant Women With a History of Bariatric Surgery, as Well as Three to Six Months After Delivery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Univ.Prof.Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PBS-1090
Record Dates: First submitted 2017-06-10; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Bariatric Surgery Candidate; Pregnancy Complications; Pregnancy Related; Glucose Metabolism Disorders
Keywords: GLP-1; Ectopic Lipids
MeSH Terms: conditions — Pregnancy Complications; Glucose Metabolism Disorders | interventions — Glucose Tolerance Test; Proton Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pregnant women with RYGB-operation (Other): Pregnant women with a history of RYGB-Operation were investigated.
  Interventions: Other: OGTT; Other: IVGTT; Other: 1H-magnetic resonance spectroscopy
- Normal weight pregnant women (Other): Normal weight pregnant women were investigated.
  Interventions: Other: OGTT; Other: IVGTT; Other: 1H-magnetic resonance spectroscopy
- Obese Pregnant women (Other): Obese pregnant women were investigated.
  Interventions: Other: OGTT; Other: IVGTT; Other: 1H-magnetic resonance spectroscopy

INTERVENTIONS:
Other: OGTT — A standardized 75g oral Glucose tolerance test was accomplished.
Other: IVGTT — For the exact assessment of Glucose metabolism in the study participants an intravenous Glucose tolerance test (IVGTT) was accomplished
Other: 1H-magnetic resonance spectroscopy — For the assessment of the ectopic lipid content in the liver, heart and the muscle a 1H-magnetic resonance spectroscopy was accomplished three to six months after delivery

SUMMARY:
In this study glucose metabolism of pregnant women with a history of bariatric surgery, obese pregnant women and normal weight pregnant women was investigated. Three to six months after delivery the assessment of Glucose metabolism was repeated and the amount of ectopic lipids in the liver, heart and muscle was measured.

DETAILED DESCRIPTION:
In this study pregnant women with a history of bariatric surgery, normal weight and obese pregnant women were invited to participate. Between the 24th and the 28th week of pregnancy an oral glucose tolerance test (OGTT), as well as an intravenous glucose tolerance test (IVGTT) was conducted. Three to six months after delivery the examinations were repeated. In addition the ectopic lipid content in the liver, heart and the muscle was measured with 1H-magnetic resonance spectroscopy and imaging three to six months post partum. The aim of this study was to compare the glucose metabolism during pregnancy between the three groups as well as to investigate the changes three to six months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a history of RYGB Operation
* normal weight pregnant women
* obese pregnant women

Exclusion Criteria:

* infectious diseases such as Hepatitis B or C, HIV, hematological diseases, acute infections, liver disease, renal disease, cancer

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2016-04-21 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Assessment of glucose metabolism using an oral Glucose tolerance test (OGTT) and an intravenous Glucose tolerance test (IVGTT) in pregnant women with a history of bariatric surgery, as well as three to six months after delivery | up to 10 months
  In this study the Glucose metabolism (including beta cell function, Insulin resistance and Insulin secretion) of pregnant women with a history of bariatric surgery was investigated with an OGTT and an IVGTT between the 24th and the 28th week of pregnancy. In Detail a measurement of the dynamic changes of Glucose, glucagon, C-peptide, Insulin and GLP-1 Levels during the OGTT and the IVGTT in pregnant women with a history of bariatric surgery was done. Three to six months after delivery the OGTT and the IVGTT were repeated and a 1H-magnetic resonance spectroscopy for the measurement of the amount of ectopic lipids in the liver, heart and the muscle was done.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Univ.Prof.Dr., Principal Investigator — Department of Internal Medicine III, Clinical Division of Endocrinology and Metabolism, Unit of Gender Medicine, Medical University of Vienna

REFERENCES:
- [Derived] Leutner M, Klimek P, Gobl C, Bozkurt L, Harreiter J, Husslein P, Eppel W, Baumgartner-Parzer S, Pacini G, Thurner S, Kautzky-Willer A. Glucagon-like peptide 1 (GLP-1) drives postprandial hyperinsulinemic hypoglycemia in pregnant women with a history of Roux-en-Y gastric bypass operation. Metabolism. 2019 Feb;91:10-17. doi: 10.1016/j.metabol.2018.10.006. Epub 2018 Nov 15. PMID 30448278